CLINICAL TRIAL: NCT03950791
Title: Single Session Pain Catastrophizing Class: Efficacy & Mechanisms for Reducing Opioid Use Among Chronic Pain Patients
Brief Title: Single Session Class to Reduce Opioid Use in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Maisa Ziadni, Clinical Instructor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 48784; K23DA047473 (NIH)
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Catastrophizing Class (Experimental): A 2-hour class that will be delivered by a clinical psychologist to participant cohorts. Didactic content includes psychoeducation about opioid use, the risk for misuse, and opioid reduction education materials.
  Interventions: Behavioral: Pain Catastrophizing Class
- Health Education (Placebo Comparator): A 2-hour in-person informational session about general health education. Participants receive a list of resources in the community.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Pain Catastrophizing Class — A 2-hour class that will be delivered by a clinical psychologist to participant cohorts. Didactic content includes psychoeducation about opioid use, the risk for misuse, and opioid reduction education materials. It will also include mind-body science as it relates to pain and PC. Participants learn how to identify catastrophizing in the moment, and how to self-treat it. During the class, participants acquire skills and develop a plan to apply the learned skills to decrease physiological hyperarousal within the context of PC. Participants also acquire skills that improve the regulation of cognition and emotion, including PC reframing and thought restructuring, and develop a plan for implementing these skills in daily life. Finally, participants develop a plan to use behaviors that modulate attention and counteract helplessness.
  Arms: Pain Catastrophizing Class
Behavioral: Health Education — Education about improving lifestyle factors to improve participants' overall health.
  Arms: Health Education

SUMMARY:
Prescription opioids are one of the most commonly used treatments for chronic pain, despite limited evidence of their efficacy and high morbidity and mortality risks. The study aims to determine the efficacy of a targeted single-session psychology class in reducing opioid use among patients with chronic pain. The information gained from this study has the potential to identify patients who achieve a meaningful reduction in opioid use and inform opioid reduction strategies.

DETAILED DESCRIPTION:
The opioid epidemic is a serious national crisis that affects public health as well as social and economic welfare, with increasing and alarming mortality rates in the United States. Consequently, there is an urgent need for effective and efficient interventions to address opioid use to prevent the risk of opioid misuse and better address it once it is established. One of the greatest predictors for increased opioid use among patients with chronic pain is pain catastrophizing (PC), defined as persistent negative cognitive and emotional responses to actual or anticipated pain. Untreated PC can lead to increased opioid use and facilitate the risk for misuse and overuse of medications, particularly when surgery and pharmacologics are the focal medical care plan. Despite critical need, there are no targeted interventions that efficiently address the key psychological factors that can amplify both pain, need for opioids, and increased risk for misuse. This project aims to address this urgent need for efficient and effective solutions. A 2-hour targeted, single-session pain catastrophizing class (PC-class) has been developed, rooted in cognitive-behavior therapy (CBT) approaches, aimed at reducing opioid use by reducing pain catastrophizing in chronic pain. This targeted, brief treatment obviates many of the existing barriers and burdens to usual comprehensive pain-CBT, such as the time required to attend 8 sessions, insurance coverage, travel costs, lack of skilled clinicians, patient attrition, and copayments. The investigators will implement a randomized controlled trial comparing the PC-class to a health education control class. Aim 1, To determine the efficacy of the PC class in reducing opioid use among patients with mixed-etiology pain conditions. Aim 2, To collect daily data that will allow the conduct of analyses on the daily experience of catastrophizing and how it relates to opioid use, as well as its dynamic response to treatment. The investigators will use this daily data to characterize the mechanistic influence of catastrophizing on opioid use both on the daily-level and prospectively. Patient outcomes will be longitudinally tracked at 1, 3, 6, and 12 months after the intervention session. This project aims to identify patients who achieve a meaningful reduction in opioid use, which will enable better characterization of treatment responders and refining opioid reduction strategies.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Diagnosis of chronic non-cancer pain (> 3 months in duration)
* Currently using prescription opioids ≥ 10mg morphine equivalent daily dose (MEDD) for ≥ 3 months;
* Ability and willingness to complete study procedures.

Exclusion Criteria:

* Open litigation regarding a medical condition
* Inability to provide informed consent and complete study procedures
* Previous experience with cognitive behavioral therapy (CBT)
* Active suicidality.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maisa Ziadni, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ziadni MS, Chen AL, Winslow T, Mackey SC, Darnall BD. Efficacy and mechanisms of a single-session behavioral medicine class among patients with chronic pain taking prescription opioids: study protocol for a randomized controlled trial. Trials. 2020 Jun 12;21(1):521. doi: 10.1186/s13063-020-04415-x. PMID 32532346

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pain Catastrophizing Class | Health Education
Started | 108 | 105
Completed | 81 | 88
Not Completed | 27 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Catastrophizing Class | Health Education | Total
Number analyzed (Participants) | 108 | 105 | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 86 | 175
  >=65 years | 19 | 19 | 38
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 86 | 83 | 169
  Male | 21 | 22 | 43
  Other | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 104 | 98 | 202
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 101 | 90 | 191
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 0 | 2 | 2
Opioid Use [Mean (Standard Deviation); unit: MME] | 133.5 (197.4) | 109.6 (163.3) | 121.7 (181.4)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use
Description: Clinically minimal reduction is defined as >15% reduction in opioid use (MEDD, which is the recommended unit of measurement in studies of opioid use)
Time Frame: baseline and 3 months
Population: Sample was comprised of participants who had available data at both baseline and primary endpoint assessments (3 months post-treatment).
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Pain Catastrophizing Class | Health Education
Number analyzed (Participants) | 84 | 91
MME | -6.7 (64.0) | -8.0 (46.8)
Statistical Analysis 1: Comparison: Pain Catastrophizing Class vs Health Education; Morphine equivalent dosage outcome variables were not normally distributed (skewness values between 4.5 and 4.8, kurtosis values between 25.7 and 30.0), which necessitated non-parametric analysis using independent-samples Mann-Whitney U Test; Test type: Superiority; p = .89, Independent-samples Mann-Whitney U — Not adjusted for multiple comparisons, p < .05 used as threshold for statistical significance; No adjustments for multiple comparisons; Mann-Whitney U = 3864, Standard Error of Mean 302.0 — Standardized Test Statistic = .139

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at baseline, pre-class assessment, and 3-, 6-, and 12-month follow-up assessments.
Arm/Group | Pain Catastrophizing Class | Health Education
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/105
Serious Adverse Events (participants affected / at risk) | 1/108 | 0/105
Other Adverse Events (participants affected / at risk) | 0/108 | 0/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pain Catastrophizing Class (N=108) | Health Education (N=105)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Not associated with the study or the intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT03950791/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT03950791/SAP_001.pdf